CLINICAL TRIAL: NCT01903278
Title: Multi-center, Randomized, Open-label, Parallel-group, Active Controlled Study for the Efficacy and Safety of Pegylated Recombinant Consensus Interferon Variant Solution for Injection in the Treatment of Chronic Hepatitis C
Brief Title: Efficacy and Safety Study of PEG-IFN-SA and Ribavirin to Treat Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Kawin Technology Share-Holding Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Cheng jun, vice president, Beijing Kawin Technology Share-Holding Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAWIN-002-2
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis c
Keywords: interferon; ribavirin; sustained virological response
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — PEG-IFN-SA; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PEG-IFN-SA /RBV T1(Genotype2,3) (Experimental): PEG-IFN-SA/RBV, 1.5μg/kg/week im and RBV 1000mg-1200mg/d po bid（BW<75kg,1000mg/d; BW≥75kg, 1200mg/d）,24 weeks
  Interventions: Drug: PEG-IFN-SA /RBV
- Pegasys /RBV C1(Genotype 2,3) (Active Comparator): Pegasys 180μg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）for 24 weeks
  Interventions: Drug: Pegasys /RBV
- PEG-IFN-SA /RBV T2(Non-genotype 2,3) (Experimental): PEG-IFN-SA 1.5μg/kg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）for 48 weeks
  Interventions: Drug: PEG-IFN-SA /RBV
- Pegasys /RBV C2(Non-genotype 2,3) (Active Comparator): Pegasys 180μg/week and RBV 1000mg-1200mg/d bid depending on body weight(BW),（BW<75kg，1000mg/d；BW≥75kg，1200mg/d）for 48 weeks
  Interventions: Drug: Pegasys /RBV

INTERVENTIONS:
Drug: PEG-IFN-SA /RBV
  Arms: PEG-IFN-SA /RBV T1(Genotype2,3); PEG-IFN-SA /RBV T2(Non-genotype 2,3)
Drug: Pegasys /RBV
  Arms: Pegasys /RBV C1(Genotype 2,3); Pegasys /RBV C2(Non-genotype 2,3)

SUMMARY:
This study is to confirm the potential effects and assess the safety of a new bio-product Pegylated Recombinant Consensus Interferon Variant Solution for Injection (PEG-IFN-SA) and Ribavirin（RBV） in the treatment of Chronic hepatitis C who have not been previously treated with Interferon.

DETAILED DESCRIPTION:
Total 720 subjects are divided into two groups and treated separately according to the HCV genotype（genotype 2,3 and non-genotype 2,3). With 2:1 ratio between experimental group and positive-control group (Peginterferon alfa-2a (Pegasys) plus RBV), 216 subjects for genotype 2,3 and 504 subjects for non-genotype2,3 will be enrolled. Accordingly, PEG-IFN-SA once weekly and RBV twice a day (bid) are given for 24 weeks and 48 weeks respectively to the HCV genotype 2,3 and the HCV non-genotype 2,3 .

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years
* Body Mass Index (BMI) 18-30
* Chronic hepatitis C , diagnosed according to Chinese guideline of Hepatitis C (year 2004)
* Detectable serum HCV-RNA by quantitative polymerase chain reaction assay and positive anti-HCV antibody
* Female subjects of childbearing age with no history of menopause and negative pregnancy test, both female and male( including their partners ) subjects were required to conduct adequate contraception since screening until the 6 months after treatment
* Volunteered to participate in this study, understood and signed an informed consent

Exclusion Criteria:

* Previous IFN treated patients
* Hepatotoxic drugs was systematically used more than two weeks within past 6 months
* Systemic therapy with potent immunomodulatory agents such as adrenocorticotropic hormone, thymosin α1, etc more than two weeks within past 6 months, not including corticosteroid nasal sprays, inhaled steroids and / or topical steroids
* Co-infection with HAV, HBV, HEV, EBV, CMV and HIV
* Evidences of hepatic decompensation, including but not limited to serum total bilirubin> 2 times the upper limit of normal (ULN); serum albumin <35g/L; prothrombin activity (PTA) <60%; ascites, upper gastrointestinal bleeding and hepatic encephalopathy; Child-Pugh score B/C grade
* Diagnosed with primary hepatocellular carcinoma or supported by evidences including but not limited to AFP> l00ng/ml, suspicious liver nodules by imaging examinations
* Liver diseases from causes other than HCV infection, including alcoholic liver disease, non-alcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis (antinuclear antibody titer higher than 1:100), hepatolenticular degeneration (Wilson's disease) and hemochromatosis, etc.
* White blood cell count <3×109/L; Neutrophil count<1.5×109/L; platelet count<90×109/L; hemoglobin below the lower limit of normal
* Serum creatinine above the ULN
* Serum creatine kinase> 3 ULN
* Diabetes mellitus or Poorly controlled Thyroid Diseases
* Poorly controlled hypertension (systolic blood pressure> 140mmHg, or diastolic blood pressure> 90 mmHg) with hypertension -related retinal lesions
* Immunodeficiency or autoimmune diseases including but not limited to inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, scleroderma, Sjogren's syndrome, autoimmune thrombocytopenia, etc.
* Psychiatric and nervous system disorders, including history of Psychiatric illness or with family history (especially depression, depressive tendencies, epilepsy and hysteria, etc.)
* Severe cardiovascular diseases (New York Heart Association functional class (NYHA) Ⅲ level and above, myocardial infarction occurred within past 6 months or PTCA performed within past 6 months, unstable angina, uncontrolled arrhythmias)
* Serious blood disorders (all kinds of anemia, hemophilia, etc.)
* Severe kidney disease (chronic kidney disease, renal insufficiency, etc.)
* Serious digestive diseases (gastrointestinal ulcers, colitis, etc.)
* Severe respiratory disease (pneumonia, chronic obstructive pulmonary disease, interstitial lung disease, etc.)
* Retinal disease (retinal exfoliation, macular hole, retinal tumors, etc.)
* Malignancies
* Function organs transplant
* Allergies or severe allergies, especially allergic to study drugs or any ingredients of the study drugs
* Evidence of alcohol or drug abuse (average alcohol consumption male> 40g / day, female> 20g / day)
* Pregnant or lactating women
* Usage of prohibition drugs in this study
* Participated in other clinical trials 3 months prior to the screening
* Unwilling to sign the informed consent and adhere to treatment requirements
* Other conditions not suitable for study judged by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
SVR (sustained virologic response) | 24 weeks after 24 or 48 weeks of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at 24 weeks after the end of SVR (sustained virologic response) defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at 24 weeks after the end of treatment

SECONDARY OUTCOMES:
RVR(rapid virologic response) | weeks 4 of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at weeks 4
cEVR (complete early virologic response) | weeks 12 of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at weeks 12
ETVR( end of treatment virologic response) | weeks 24 of study therapy for genotype 2,3, and weeks 48 of study therapy for non-genotype 2,3
  defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at the end of treatment
eRVR ( extended rapid virologic response) | weeks 4 and 12 of study therapy
  defined as the proportion of patients who had undetectable plasma HCV RNA (HCV RNA < 15 IU/mL) at weeks 4 and 12
No-responses | weeks 12 or weeks 24 of study therapy
  defined as the proportion of patients who had less than a <2 log IU/ml plasma HCV RNA decline at weeks 12 or had detectable plasma HCV RNA at weeks 24
Breakthrough | weeks 12, 24 of study therapy for genotype 2,3, and weeks 12, 24 and 48 of study therapy for non-genotype 2,3
  defined as the proportion of patients who had detectable plasma HCV RNA at any point during treatment after virological response( undetectable plasma HCV RNA)
Relapse | 12 and 24 weeks after 24 or 48 weeks of study therapy
  defined as the proportion of patients who had undetectable HCV RNA at the end of treatment, but reappearance of HCV RNA after the then

CONTACTS AND LOCATIONS:
Overall Officials: Cheng jun, MD, PhD, Principal Investigator — Beijing Ditan Hospital
Locations (41):
- China (41):
  - First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical Unbiversity, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Union hospital, Tongji Medical College Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Jiangsu province hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital (Yanbian Hospital), Yanji, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - First Affiliated Hospital Of Medical College of Xian Jiaotong University, Xi'an, Shaanxi
  - Second Affiliated Hospital Of Medical College of Xian Jiaotong University, Xi'an, Shaanxi
  - Tangdu Hospital，Fourth Military Medical University, Xi'an, Shaanxi
  - Jinan Infectious Disease Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong university, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Science ＆Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - 302 Military Hospital of China, Beijing
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, capital Medical University, Beijing
  - General Hospital of Beijing Military Region, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Chongqing Southwest Hospital, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Shanghai Public Health Clinical Center, Shanghai
  - Tianjin Infectious Disease Hospital, Tianjin